

### **Master Informed Consent Form**

[Investigator name]

[Investigator address or affiliation]

[Investigator telephone number]

[IRB/IEC name]

**Study Title:** A First-in-Human, Open Label, Phase I/II Study to Evaluate the Safety,

Tolerability and Pharmacokinetics of HH2710 in Patients with

**Advanced Tumors** 

**Protocol Number:** HH2710-G101

**Sponsor:** Haihe Biopharma Co., Ltd.

Name of Investigator or Other Person Administering Consent: [Name of Investigator or other person]

### **Important**

This informed consent ("permission") form may contain words that you do not understand. Please ask the study doctor or the study staff to explain any words or information that is not clear to you.

Joining a study is an important decision. You should ask the study team any questions you may have about the study and this informed consent form before making a decision to participate.

Also, you may have your primary doctor call the study doctor to ask any questions he/she feels are necessary to evaluate the study and your possible participation in it.

You may take home an unsigned copy of this informed consent form to think about it or discuss it with family or friends before making your decision to take part in the study.

This document is confidential.

Subject Initials: \_\_\_\_\_Date: Master ICF Version Number: 3.0 Date: 22-Mar-2022 Controlled Document ID: **4106A**, Effective Date: 30-Apr-2018

<sup>&</sup>quot;Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inventive Health group of companies"

### Why is this study being done?

Haihe Biopharma has begun a study of an investigational drug (also known as the "study drug") called HH2710 as a possible treatment for advanced tumors. An investigational drug is one that has not been approved by the United States (US) Food and Drug Administration (FDA). You are being asked to take part in this study because you have been diagnosed with advanced tumors. If you do not want to take part in the study, your decision will be respected. This study involves research.

Your participation in this study is voluntary. If you decide not to take part in this study, you can continue with your current medical care.

The main purpose of this study is to learn how well the study drug works and how safe the study drug is.

### How many people will take part in this study?

This study will be conducted in 2 Phases: Phase I (also known as a "first-in-humans" study) and Phase II (the next phase of the study to determine whether the drug has any biological activity or effect). This study has 3 parts including Phase I dose escalation (to establish the maximum tolerated dose [the highest dose that does not cause unwanted side effects]), Phase I dose expansion (additional people are enrolled to collect more information), and Phase II dose extension (further effect of study drug will be studied in this phase).

A total of approximately 58 people will be enrolled in Phase I dose escalation part, an additional 10 people per dose cohort will be enrolled in Phase I dose expansion part; the total number of people in this part will depend upon number of doses to be studied. Approximately 108 people will be enrolled in Phase II dose extension part of the study. You will participate in only one phase of the study.

### How long will my participation in this study last?

Your participation in this study will last until you or your doctor decides your participation should end, or progression of your disease (your tumor gets worse), or the Sponsor stops the study, whichever comes first. You will need to visit the research site for the screening visit, 3 times each during Cycle 1 and Cycle 2, and then whenever dictated by your health or the study doctor, but at least once every 2 cycles of a 21-day cycle from Cycle 3, then at the end of treatment visit, safety follow-up visit, and disease progress follow-up visit. You will be contacted by telephone for survival follow-up visit.

#### What will happen during this study?

The study is divided into 2 phases. During this study (both the phases), there is a screening visit, a baseline visit, 1 or more treatment cycles, an end of treatment visit, a safety follow-up visit, a

This document is confidential.

<sup>&</sup>quot;Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inventive Health group of companies"

disease progress follow-up visit, and a survival follow-up visit. You might have only 1 treatment cycle during this study, or you might have 2 or more treatment cycles if the study doctor determines that you meet the requirements for additional treatment cycles.

During each study period, you will have 1 or more visits with the study doctor at the center. The screening visit and the treatment period visits will last about 3 to 4 hours, and all other visits will last about 1 to 2 hours.

Before any study-related tests and procedures can be done, you will be asked to read and sign this informed consent form. After you sign this informed consent form, the study will begin with a screening visit. The purpose of the screening visit is to determine if you meet the requirements to take part in this study. If you do not meet the requirements, the study doctor will explain why and will discuss with you other treatment options.

**Phase I**: The first 3 patients will receive an HH2710 capsule 1 time on the first day, followed by twice every day orally (by mouth) during a 21-day cycle from the second day. The fourth and later patients will take study drug orally every day during a 21-day cycle from the first day following the dosing schedule and instructions, which is very important. You are required to fast for about 2 hours before and after taking the study drug. All the patients who will take part in this phase will receive 1 of the doses as described in the table below. The dose level and frequency will be assigned to you by your study doctor, depending upon when you will enter the study.

### The dosing and treatment schedule:

| Dose<br>Level | Dose of HH2710 | Patient | Study Drug form and route of administration | Dosing Frequency |
|---|---|---|---|---|
| Level 1 | 25 mg | 3 | Capsules for oral use | QD at C1D1, then BID from C1D2 (21 days/cycle) |
| Level 2 | 50 mg | 3 | Capsules for oral use | BID (21 days/cycle) |
| Level 3 | 100 mg | 3+N# | Capsules for oral use | BID (21 days/cycle) |
| Level 4 | 300 mg | 3+N# | Capsules for oral use | QD (21 days/cycle) |
| Level 5 | 400 mg<br>(Total daily dose*) | 3+N | Capsules for oral use | QD/BID (21 days/cycle) |
| Level 6 | 600 mg<br>(Total daily dose*) | 3+N | Capsules for oral use | QD/BID (21 days/cycle) |
| Level 7 | 800 mg<br>(Total daily dose*) | 3+N | Capsules for oral use | QD/BID (21 days/cycle) |

Abbreviations: QD = once daily; BID = twice daily; C1D1 = Cycle 1 Day 1; C1D2 = Cycle 2 Day 2.

This document is confidential.

<sup>#:</sup> The number of subjects enrolled in each dose is specified by the Bayesian optimal interval rules;

<sup>\*:</sup> Proposed daily dose is the total dose each day with QD or BID dose frequency.

Dosing frequency and dose level may be adjusted on the basis of available pharmacokinetic data and safety.

<sup>&</sup>quot;Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inventive Health group of companies"

**Phase II**: The recommended dose level and frequency for Phase II will be decided based on Phase I results. All patients enrolled in this phase will take the study drug orally once daily (QD)/twice daily (BID) during a 21-day cycle. You will be enrolled in one of the 4 cohorts depending upon your disease type. It is very important that you follow the dosing schedule and instructions. You are required to fast for about 2 hours before and after taking the study drug.

### **Study Procedures and Assessments**

This is a description of the procedures and assessments that will be performed during the study, including the prescreening and screening visits, is shown below. In addition to the visits described below, the study doctor may ask you to come in for extra visits, if necessary, for your safety.

### Molecular Screening Visit

You will be asked to provide molecular screening consent before any other study-related procedures and assessments. Please read the information below for more details.

Consent for Genetic Analysis: An archived tumor tissue or slices (means previously collected and stored) or fresh tumor biopsy sample will be collected for molecular screening. You will be asked to provide your consent on the "Molecular Screening Informed Consent (Biomarker ICF)" to take part in this study. The biomarker samples (samples of substances in your body that can measure the presence of disease or the effects of treatment) will be used to study the biology (eg, DNA, RNA, proteins, and metabolites) to understand how HH2710 works and to learn about advanced tumors.

Participation in this testing is mandatory in Phase II stage. If you do not want your genotyping sample to be used in this molecular screening, you cannot take part in the main study. If you agree to the genotyping testing, you will be provided with separate informed consent document (Biomarker ICF) to sign. As for Phase I dose expansion stage, you are required to provide the local laboratory test results of MAPK pathway gene alteration status to determine the eligibility of patient participating in clinical screening procedure. Your study doctor will tell you which phase you will be in if you are willing to join the study.

### Screening Visit

The study doctor will perform the following examinations and tests to determine if you should take part in the study:

- 1. You will be asked about your health and the medicines that you have taken or are currently taking, and the medical procedures that you have had.
- 2. You will be asked about your cancer diagnosis and treatment history.
- 3. Your birth date, sex, and race, per national regulations, will be recorded.
- 4. You will be assessed for your disease-related signs and symptoms.

"Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inventive Health group of companies"

This document is confidential.

Subject Initials: \_\_\_\_\_Date: Master ICF Version Number: 2.2 Date: 17-Jul-2021 Controlled Document ID: 4106A, Effective Date: 30-Apr-2018

- 5. The study doctor will perform a physical examination to check your overall health, including height and weight.
- 6. Your blood pressure, heart rate, respiratory rate, and body temperature will be measured.
- 7. An electrocardiogram (ECG) will be done. This is a test that measures the electrical activity of the heart. A technician will place patches on your chest that will be connected by wires to a machine. The machine will record the electrical activity of your heart.
- 8. The study doctor will examine you and will also assess how your cancer affects your daily activities (Eastern Cooperative Oncology Group [ECOG] performance status).
- 9. The study doctor will examine your eyes.
- 10. A urine sample (about ½ cup) will be taken to check your overall health.
- 11. Echocardiogram (ECHO; a soundwave test of your heart) or multigated acquisition (MUGA; video test of your heart) scan will be done
- 12. Tumor measurements including computed tomography (CT) or magnetic resonance imaging (MRI) scans.
- 13. Tumor tissue may be collected by biopsy for central histological review (ie, by microscopy) of your disease and biomarker analyses, which depends on the study phase you participate in.
- 14. Blood samples will be collected for the following laboratory tests. Approximately 7 ½ teaspoons or 37 mL of blood will be taken from your arm using a needle.
  - Safety laboratory tests will be done to check your overall health.
  - Cardiac function tests will be done to measure troponin (a protein that controls muscle contraction) levels in your blood.
  - If you are a woman who is able to have children, your blood will be tested to see if you are pregnant. The results of the pregnancy test must be negative in order for you to participate in this study.
  - Tests will be done to screen for certain viruses (including human immunodeficiency) virus and hepatitis B and C viruses). If your test result is positive and you have given or received blood, blood products, organs, or tissues, the Public Health Department will be notified as required by law. These tests are mandatory. If you decline these tests, you will not be allowed to participate in the study.
- 15. The study doctor will review any side effects experienced after signing this informed consent form.

#### **Treatment Period**

The study doctor or the study doctor's staff will perform the following tests and procedures. You will be asked to visit the study site 3 times each during Cycle 1 (baseline [Day 1], Day 8, and Day 15) and Cycle 2 (Day 22, Day 29, and Day 36) and then on the 1st day of every 2 cycles

This document is confidential.

Subject Initials: Master ICF Version Number: 2.2 Date: 17-Jul-2021 Controlled Document ID: 4106A, Effective Date: 30-Apr-2018

<sup>&</sup>quot;Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inventive Health group of companies'

Principal Investigator: <PI name>; Site No.: <site #>

starting from Cycle 3 (Day 43). The study staff will explain to you in detail about study site visits.

- 1. You will be asked about your cancer diagnosis and treatment history.
- 2. You will be assessed for your disease-related signs and symptoms.
- 3. You will be asked about your health and the medicines that you have taken or are currently taking, and the medical procedures that you have had.
- 4. The study doctor will perform a physical examination to check your overall health and weight; after the screening visit, the physical examination will be performed if the study doctor believes you need it. Also, the study doctor will examine your eyes, if needed.
- 5. Your blood pressure, heart rate, respiratory rate, and body temperature will be measured.
- 6. The study doctor will examine you and will assess how your cancer affects your daily activities (ECOG performance status).
- 7. The study doctor will examine your eyes.
- 8. If you are a woman who is able to have children, your blood will be collected and tested to see if you are pregnant at the baseline. After the baseline, your urine pregnant result is also accepted during the treatment period.
- 9. Study drug will be provided at each study visit.
- 10. Study drug should be administered continuously, according to dose schedule.
- 11. Tumor measurements including CT or MRI scans (every 2 cycles, approximately every 6 weeks  $\pm 7$  days).
- 12. An ECG will be done at each study visit. (Note: ECGs will be obtained prior to dosing and 1, 3, 4, and 8 hours after dosing on Cycle 1 Day 1 and Cycle 2 Day 1).
- 13. An ECHO or MUGA scan should be measured at your study doctor's discretion if there are signs or symptoms of cardiotoxicity (damage to your heart) during the study.
- 14. A urine sample (about 1/2 cup) will be taken to check your overall health (may not be performed at the Baseline visit, based on your doctor's decision).
- 15. Blood samples will be collected for the laboratory tests listed below. Approximately 7 ½ teaspoons or 37 mL of blood will be taken from your arm using a needle.
  - Safety laboratory tests will be done to check your overall health (may not be performed at Baseline visit based on your doctor's decision).
  - If you are a woman who is able to have children, your blood will be tested to confirm if you are pregnant when the urine pregnancy test is positive.
- 16. The following blood tests will be performed during Phase I dose escalation stage only on Day 1, Day 2, Day 7, Day 10, Day 15, and Day 16 of Cycle 1; on Day 1 of Cycles 2, 3, 5, 7, and 9; and during Phase I dose expansion stage and Phase II dose extension on Day 1, Day 2, Day 15 and Day 16 of Cycle 1 (only pharmacokinetic samples):

This document is confidential.

Subject Initials: Master ICF Version Number: 2.2 Date: 17-Jul-2021 Controlled Document ID: 4106A, Effective Date: 30-Apr-2018

<sup>&</sup>quot;Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inventive Health group of companies'

Principal Investigator: <PI name>; Site No.: <site #>

• Pharmacokinetic (PK) tests will be done to look at how your body metabolizes (breaks down) the study drug. The blood samples will be taken before and after the study drug administration.

- 17. The following blood tests will be performed during Phase I only at Day 1 and Day 15 of Cycle 1 (only conducted in sites that are capable of sample collection and processing for Pharmacodynamic samples):
  - Pharmacodynamic (PD) tests for certain blood components called biomarkers (markers of drug response including phosphorylation of ribosomal S6 kinase [pRSK and total RSK]) will be done to learn more about how the study drug affects your body and to better understand how the study drug works.
- 18. You will be asked to return all the unused study drug at each study site visit.
- 19. Study drug compliance will be assessed by capsule count at each visit.
- 20. Review of side effects experienced since your previous study visit.

# End of Treatment/Early Discontinuation Visit

For all patients who leave the study before study completion, the study doctor's staff will perform the following tests and procedures within 7 days of the last dose:

- 1. You will be asked about your cancer diagnosis and treatment history.
- 2. You will be assessed for your disease-related signs and symptoms.
- 3. You will be asked about your health and the medicines that you have taken or are currently taking, and the medical procedures that you have had.
- 4. The study doctor will perform a physical examination to check your overall health, including weight.
- 5. Your blood pressure, heart rate, respiratory rate, and body temperature will be measured.
- 6. The study doctor will examine you and will also assess how your cancer affects your daily activities (ECOG performance status).
- 7. The study doctor will examine your eyes.
- 8. A urine sample (about 1/2 cup) will be taken to check your overall health based on your doctor's decision.
- 9. If you are a woman who is able to have children, your urine or blood will be tested to see if you are pregnant.
- 10. Tumor measurements including CT or MRI scans.
- 11. An ECG will be done.
- 12. Blood samples will be collected for the following laboratory tests. Approximately 7 ½ teaspoons or 37 mL of blood will be taken from your arm using a needle.

This document is confidential.

Subject Initials: \_\_\_\_\_Date: Master ICF Version Number: 2.2 Date: 17-Jul-2021 Controlled Document ID: 4106A, Effective Date: 30-Apr-2018

<sup>&</sup>quot;Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inventive Health group of companies"

Principal Investigator: <PI name>; Site No.: <site #>

- Safety laboratory tests will be done to check your overall health.
- 13. You will be asked to return all the unused study drug.
- 14. Study drug compliance will be assessed by capsule count.
- 15. Review of side effects experienced since your previous study visit.

### Follow-Up Period

### Safety Follow-Up Visit

A safety follow-up visit will be scheduled within 30 days (+ 7 days) after the last dose of study drug. At this visit, the study doctor or the study doctor's staff will perform the following tests and procedures:

- 1. You will be asked about the medicines that you have taken or are currently taking.
- 2. An ECG will be done.
- 3. A urine sample (about  $\frac{1}{2}$  cup) will be taken to check your overall health.
- 4. Blood samples will be collected for the following laboratory tests. Approximately 7 ½ teaspoons or 37 mL of blood will be taken from your arm using a needle.
  - Safety laboratory tests will be done to check your overall health, which including blood routine, blood biochemistry, thyroid function, and coagulation as protocol required.
- 5. Echocardiogram (ECHO; a soundwave test of your heart) or multigated acquisition (MUGA; video test of your heart) scan will be done.
- 6. Review of side effects experienced since your previous study visit.
- 7. You will be asked about the new treatment for your disease and survival condition i.e. your present health.

### Follow-Up of Progressive Disease

A follow-up visit to check progression of your disease will be scheduled once every 6 weeks after the last dose of study drug. At this visit, the study doctor or the study doctor's staff will perform the following tests and procedures:

- 1. Tumor measurements including CT or MRI scans.
- 2. You will be asked about the new treatment for your disease and survival condition i.e. your present health.

<sup>&</sup>quot;Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inventive Health group of companies"

Principal Investigator: <PI name>; Site No.: <site #>

### **Survival Follow-Up**

All patients who discontinued from study drug for any reason will be contacted every 3 months by telephone from the time of worsening of their disease or starting a new treatment to 1 year in order to inquire about their status.

### What do I have to do?

During the study, you will have the following responsibilities:

- Tell your study doctor if you have any allergies, including drug allergies. If you are unsure, ask your primary doctor.
- Attend all scheduled visits.
- Take the study drug as directed.
- Return any unused study drug and containers as instructed by the study staff.
- Follow the study doctor's instructions about whether you may continue to take your regular prescribed medications or over-the-counter medicines during the study period.
- Tell the study doctor of any changes to your current medications, illnesses or injuries, unexpected or troublesome side effects, or problems that occur during the study.
- Tell the study doctor if you plan to have an elective surgery or any other medical treatment or procedure.
- You should not perform activities requiring mental alertness, judgment, or physical coordination such as driving or operating machinery, or doing anything that requires you to be alert, unless you feel secure and safe to do so.
- You should continue to make regular visits to your primary doctor or any other special doctors whom you were seeing before starting the study, because being in the study does not replace regular medical care.
- Make sure that the study drug is kept out of the reach of children and people who have a limited capacity to read or understand. You are the only person who should take the study drug.
- Contact the study doctor if you find you have any questions about the study after you sign this form.
- You and/or your partner must use a reliable form of contraception during the study. If you or your partner becomes pregnant while you are in the study, be sure to tell the study doctor as soon as possible.

### What are the benefits of being in this study?

There is no guarantee that you will receive any benefits. However, you will be helping others by contributing to medical research. Additionally, you may experience some benefits, for example, your symptoms can improve and your tumor might shrink.

<sup>&</sup>quot;Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inventive Health group of companies'

### What are the risks and possible discomforts?

If you choose to take part in this study, there are risks that:

- You may lose time at work or home and spend more time in the hospital or doctor's office than usual.
- You may be asked sensitive or private questions which you normally do not discuss.

The drug used in this study may affect the function of other organs, such as your liver, kidneys, heart, and blood. The study doctor will be testing your blood and will inform you if changes occur that may affect your health.

There is also a risk that you could have side effects from the study drug and the study approach.

Here are important points about side effects:

- The study doctors do not know who will or will not have side effects.
- Some side effects may go away soon, some may last a long time, or some may never go away.
- Some side effects may interfere with your ability to have children.
- Some side effects may be serious and may even result in death.
- Tell the study doctor if you notice or feel anything different so they can see if you are having a side effect.
- The study doctor may be able to treat some side effects.
- The study doctor may adjust the study drugs to try to reduce side effects.

The study drug has not been used in humans before, so the side effects are unknown at this time. However, based on its mode of action (the way the drug affects the body) and studies in animals, its side effects are thought to be similar to other drugs of same target class described below. There might be other side effects that researchers do not yet know. The common and possible side effects are listed in the following tables.

| Common Side Effects | diarrhea, nausea, vomiting, decreased appetite, abdominal (belly) pain, impaired gastric emptying (stomach doesn't empty food as quickly as it should), rash, pruritus (itchy skin), alopecia (hair loss), fatigue, chills, increased serum bilirubin (blood levels of a liver compound), increased blood urea nitrogen (a waste product from the liver), increased blood creatinine (a waste product from muscles), anemia (low level of red blood cells), and altered taste |
|---|---|
| Potentially Severe Side Effects | retinal vein occlusion (blockage of small veins that carry blood away from the retina [part of your eye]), |

<sup>&</sup>quot;Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inventive Health group of companies"

This document is confidential.

Subject Initials: \_\_\_\_\_Date: Master ICF Version Number: 2.2 Date: 17-Jul-2021 Controlled Document ID: 4106A, Effective Date: 30-Apr-2018

Principal Investigator: <PI name>; Site No.: <site #>

| which<br>failur | papathy (damage to the blood vessels in the eye<br>in may cause vision problems), acute renal (kidney)<br>e, increased creatine phosphokinase (a protein that<br>chemical changes happen in your body) |
|---|---|
|---|---|

Let your study doctor know of any questions you have about possible side effects.

### **Pregnancy/Birth Control**

Because the effect of study drug on unborn babies is not known, you should not become pregnant, breastfeed, or father a baby while in this study.

#### Women

Taking the study drug may involve unknown risks to a pregnant woman, an embryo, fetus (unborn baby), or breastfeeding infant. Therefore, if you are pregnant, planning to become pregnant, or are breastfeeding a child, you cannot take part in this study.

Before entering the study, a pregnancy test will be done for all women who are able to become pregnant. This test might not detect an early pregnancy. Pregnancy tests will be repeated during the study.

The only certain way not to become pregnant is to not have sex. If you choose to have sex during the study, you must use an effective method of birth control while you are taking part in this study and for 6 months after you finish the study treatment. If you are already using a method of birth control, the study doctor or study staff will discuss with you whether your current method of birth control is acceptable for use during this study. Methods of effective birth control include surgery, hormonal contraceptive, patch, vaginal ring, intrauterine device, or double physical barrier such as condoms plus diaphragm.

If during the study you become pregnant, you should tell the study doctor as soon as possible. The study drug will be stopped, and your involvement in this study will end.

### Men

Male subjects should be surgically sterile or compliant with a highly effective contraceptive method during the study and for a minimum of 6 months after you finish the study treatment. These may include surgery or a physical barrier such as a condom.

The Sponsor may like to receive updates on the progress of the pregnancy and its outcome. If you agree to this, you will be asked to sign a separate informed consent.

### What if there are new findings?

"Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inventive Health group of companies"

This document is confidential.

Principal Investigator: <PI name>; Site No.: <site #>

If new findings that would affect your safety and willingness to participate in the study are identified while you are in the study, you will be told as soon as possible, so you can decide whether to leave the study or continue. If you continue, you will be required to sign a new informed consent form.

### What other options are available if I do not take part in this study?

You do not have to take part in the study to treat your advanced tumor. By participating in this study, you may be foregoing effective therapies that may include FDA-approved therapies which may shrink tumor, delay progression of cancer, or provide symptom relief, if those therapies are available in your country. There are other options of therapies, such as immunotherapy, chemotherapy, dabrafenib, trametinib, vemurafenib, cobimetinib, encorafenib, and binimetinib.

Your primary doctor or the study doctor can answer any questions that you have about other treatments.

You should also contact your primary doctor to ask about other research currently being done in the treatment of advanced tumor.

### Who is paying for this study?

Haihe Biopharma is funding this study. The study doctor will be paid for his/her work in this study.

### What are the costs?

The study drug will be given at no cost to you, and you will not be charged for any study doctor visits, laboratory work, tests, or procedures that are needed for the study.

### Will I be paid for being in the study?

You will receive no payment for taking part in this study. However you may be reimbursed for any reasonable travel, parking, meals, and other expenses associated with the research project visit, upon approval from the Sponsor, Haihe Biopharma.

### What if I get sick or hurt?

If you require medical treatment for an illness or injury that is a direct result of taking the study drug, Haihe Biopharma will pay for reasonable and routine costs of such treatments if the following conditions are met:

- The illness or injury was a result of taking part in the study.
- The cost of treatment or any part of the costs is not covered by any other health insurance, government health program, or other institutions providing coverage for health care.

<sup>&</sup>quot;Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inventive Health group of companies"

### Can I leave the study after it has begun?

Yes. Taking part in this study is voluntary, and you can leave the study at any time for any reason. There will also not be any penalty or loss of benefits to which you are entitled at this site if you decide not to take part or if you decide to leave the study.

If you decide to leave the study, you should contact the study doctor who will explain the safest way to end participation, which may involve the completion of some final tests and examinations. You should also contact your primary doctor so he or she can provide you with the best course of continuing care.

The study doctor or Haihe Biopharma can remove you from the study, without your permission, for some reasons. Possible reasons for doing so include the following:

- Any change in your medical condition that might make continuation in the study harmful to you
- Your failure to follow the study doctor's instructions
- Discovery that you do not meet the study requirements
- Cancellation of the study
- Administrative purposes: For example, insufficient drug supply or site closing etc.

### What will happen to the samples that I provide?

The blood samples that you give will be used only for specific tests that are needed for this study. Your samples will be destroyed as soon as possible after those specific tests are completed. Your samples will be tested and destroyed according to the standard procedures of the laboratory.

### What happens when this study stops?

When the study stops, you will be under the care of your primary doctor who will decide the best way to treat your disease. The study drug will no longer be available to you.

You have the right to be informed of the overall results of the study.

### Will my records be kept private?

To participate in this study, you must read and sign the Privacy Notice at the end of this form (see Appendix 1).

### What if I have a question or concern?

You should feel free to ask questions about the study and your rights as a subject before, during, and after the study.

<sup>&</sup>quot;Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inventive Health group of companies"

Informed Consent Form

Sponsor: Haihe Biopharma Co., Ltd.; Protocol No.: HH2710-G101

Principal Investigator: <PI name>; Site No.: <site #>

### Whom can I call?

If you have any questions about this study or if at any time you believe that you have a research-related injury or a reaction to the study drug, you should contact <insert study doctor's name> by telephone at <insert his/her telephone number>.

If you have any questions regarding your rights as a research subject, you may contact <insert IRB/IEC name> by telephone at <insert IRB/IEC telephone number>.

### **Important**

Do not sign this informed consent form unless you have had a chance to ask questions and have received satisfactory answers to all of your questions.

Signing your name to this informed consent form means that you voluntarily agree to take part in this study.

This agreement can be withdrawn at any time; although, data collected up to that point is legally allowed to be used.

<sup>&</sup>quot;Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inventive Health group of companies"

Informed Consent Form


Principal Investigator: <PI name>; Site No.: <site #>

# **Consent to Participate**

By signing this informed consent form, I agree to the following:

- I have read, and I understand this informed consent form.
- I have been given the chance to ask any questions that I had about the study, and all questions that I asked were answered to my satisfaction.
- I understand the risks of taking part in this study as described in this informed consent form.
- I understand that there is no guarantee that I will receive any benefits from taking part in this study.
- I freely consent to be treated with drug under the study doctor's care.
- I confirm that all information that I have given about my medical history is correct to the best of my knowledge.
- I understand that I am free to withdraw from the study at any time for any reason. I will tell the study doctor if I decide to withdraw so that my participation may end in an orderly manner, and my future care can be discussed.
- I understand that I will be told of any new information that might relate to my willingness to continue in the study.
- I will tell the study doctor if I have any physical or psychiatric ("mental health") symptoms or problems.
- I understand that I will receive a signed and dated copy of this informed consent form for my records.

My consent to participate in this study does not take away any legal rights in the case of negligence (carelessness) or other legal fault of anyone who is involved with this study.

| Name of participant (print) | |
|---|---|
| Signature of participant | Date (dd/Mmm/yyyy) |
| Signature of study doctor or person administering consent | Date (dd/Mmm/yyyy) |

This document is confidential.

Subject Initials: \_\_\_\_\_Date: Master ICF Version Number: 2.2 Date: 17-Jul-2021 Controlled Document ID: 4106A, Effective Date: 30-Apr-2018

<sup>&</sup>quot;Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inventive Health group of companies"

# **Appendix 1: Privacy Notice**

**Identification of Data Controller:** During the study, the Sponsor will direct the collection and use of your personal information (data) needed for the study. The Sponsor is the data controller of your personal data under applicable data protection laws. You can contact the Sponsor at:

Ms. Xianqing Hu

Haihe Biopharma Co., Ltd.

No. 865 Zuchongzhi road, Pudong New Area, Shanghai, China

Tel: +86 21 20568888

The study center may also be considered as a data controller of your personal data under applicable data protection laws. You may contact the study doctor using the contact information for the study doctor on the first page of this informed consent form.

If you have any questions or would like to see the data collected about you for this study, you should contact the study doctor.

**Data to be Collected and Processed:** The study staff will collect data about you for the study. This data may include your name or initials, date of birth, gender, contact details, and information needed for payment processing. In addition, the following sensitive personal data about you may be collected: health, race, genetic information.

How Your Personal Data Will be Used: The personal data collected about you will be recorded in your study file by the study staff to run the study and to monitor your safety as a participant. Your personal data may be processed on a computer and/or on paper. The collection of this data is necessary to conduct the study and comply with applicable laws. You will not be able to participate in the study if you fail or refuse to provide your information.

There are laws about the recording, forwarding, storage, and analysis of your personal data, including sensitive personal data. These laws require your voluntary and explicit consent before you participate in the study. If you do not consent to the collection and use of your personal information, you will not be able to be in the study.

Results of this study may be presented at meetings or in publications; however, your identity will never be shared. Your personal data will not be used for any direct marketing purposes.

If information regarding a communicable disease is collected, the information may be shared with a public health authority that is authorized by law to collect or receive such information for the purpose of preventing or controlling disease, injury, or disability, and conducting public health surveillance, investigations, or interventions.

This document is confidential.

Subject Initials: Master ICF Version Number: 2.2 Date: 17-Jul-2021 Controlled Document ID: 4106A, Effective Date: 30-Apr-2018

<sup>&</sup>quot;Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inventive Health group of companies'

Principal Investigator: <PI name>; Site No.: <site #>

**Storage of Your Personal Data:** According to legal requirements, your personal data will be stored in the study databases and/or paper files for at least 15 years after the study ends, as required by applicable laws.

Transferring the Personal Data to a Third Party: To keep your identity private, all data that is sent or provided outside of the study center will show only a coded identification number instead of your name. Only the study doctor and authorized personnel will be able to connect this code to your name. They will use a list that will be kept in a secure place to link this code to your name in case of an emergency. The coded data from the study showing your involvement (including uncoded personal information) will be provided to the Sponsor and other individuals and/or companies that act on the Sponsor's behalf, including Syneos Health. Also, your medical records (including uncoded personal data) may be reviewed by the Sponsor and other individuals and/or companies that act on the Sponsor's behalf, including Syneos Health; government agencies in countries where the study drug may be considered for approval (such as the US FDA); [IRB/IEC name], a group that reviews and approves studies; and independent auditors for the purposes of confirming your participation in the study, monitoring your safety during the study, and monitoring the conduct of the study. Further, your personal information may be disclosed in response to lawful requests by public authorities, including those to meet national security or law enforcement requirements.

If your personal data is shared with other companies that are located outside of the country where you live, the Sponsor will make sure your data is protected as required by your country's data protection laws. Some of these other companies may be located in countries whose data protection and privacy laws may be less strict than in your own country, including the United States and \_\_\_\_\_\_. You may contact the study doctor to get more information about the precautions used to protect your personal data outside of your country. You may also ask the study doctor for a copy of those precautions.

With your permission, the study doctor will tell your primary doctor about your role in this study.

A description of this clinical trial will be available on http://www.clinicaltrials.gov as required by US law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

Your Rights as a Data Subject: You have the right to access and correct the data collected about you during the study and submit any questions or concerns about the collection or processing of your personal data; however, this access is suspended until after the study has ended. Your rights will be reinstated at the conclusion of the study.

You have the right to withdraw your consent for the processing of your personal data at any time. You must withdraw your consent by writing to the study doctor. However, data collected before

This document is confidential.

<sup>&</sup>quot;Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inventive Health group of companies"

Informed Consent Form


Principal Investigator: <PI name>; Site No.: <site #>

you remove your consent is still legally allowed to be used. If you withdraw your consent, you will no longer be able to take part in the study.

### Consent Language

### Consent to the Collection, Processing, and Use of Personal Data

By signing below, I agree that:

- (1) My personal data, including sensitive personal data, can be collected, used, and archived for purposes of carrying out the study as described in this Privacy Notice;
- (2) My personal data, including sensitive personal data, can be transferred to and shared with other companies both within and outside of the European Economic Area (EEA), including to countries that may not have the same level of data protection as the EEA, as described in the Privacy Notice;

This consent is valid unless you change your mind and provide a written notice to the study doctor. You will receive a signed and dated copy of this Privacy Notice.

| Name of participant (print) | <u> </u> |
|-----------------------------|--------------------|
| | <u> </u> |
| Signature of participant | Date (dd/Mmm/yyyy) |

This document is confidential.

Subject Initials: \_\_\_\_\_Date: Master ICF Version Number: 2.2 Date: 17-Jul-2021 Controlled Document ID: 4106A, Effective Date: 30-Apr-2018

<sup>&</sup>quot;Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inventive Health group of companies"



[Investigator name]

[Investigator address or affiliation]

[Investigator telephone number]

[IRB/IEC name]

**Study Title:** A First-in-Human, Open Label, Phase I/II Study to Evaluate the Safety,

Tolerability and Pharmacokinetics of HH2710 in Patients with Advanced Tumors

Protocol No.: HH2710-G101

**Sponsor:** Haihe Biopharma Co., Ltd.

Name of Doctor or Other Person Administering Consent: [Name of doctor or other person]

# **Introduction and Purpose of Genetic Analysis**

You are a participant in a clinical study with HH2710 being investigated for the treatment of advanced tumors, and you are being asked if you would like to take part in a genetic analysis called as molecular screening. Before you decide, we would like you to understand why the research is being done and what it would involve for you. One of the study staff will go through this informed consent with you and answer any questions you may have. Talk to others about the study if you wish.

Your participation in the molecular screening is mandatory in Phase II stage. In case you refuse to participate in this analysis, you cannot participate in the main study.

If you agree to participate, you will be asked to sign the molecular screening informed consent form at the end of this document before your tumor biopsy or tissue samples are collected.

### Purpose and background

Your genetic data consist of genes and other biological and chemical processes, structures, and sequences (for example, DNA, RNA, chromosomes, genes, proteins, and metabolites), all of which are in your blood and body tissues. These genetic data make you different from anyone else. Some genetic data control things like the color of your hair or eyes. Other genetic data might make you more likely to get certain diseases or affect whether a drug helps you and/or gives you side effects. Genetic tests might be used to sequence your DNA, RNA, chromosomes,

<sup>&</sup>quot;Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inVentiv Health group of companies"


Principal Investigator: <PI name>; Site No.: <site #>

and genes, but analyses of genetic tests will be limited only to results that might relate to the study drug, the disease, and your medical conditions.

Mitogen-activated protein kinase (MAPK) is a type of protein kinase that is specific to the amino acids serine and threonine, which are important molecules in transmitting signals from the surface of a cell to its nucleus (center). They regulate cell functions including proliferation (growth and increase), gene expression (the process of gene information becoming a useful product), differentiation (changing from one cell type to another), mitosis (division of cells), cell survival, and apoptosis (cell death).

For the Phase I does escalation, determination of the MAPK pathway gene alteration status is not required, but information will be collected and documented if available. For the Phase I expansion stage, local laboratory test results of MAPK pathway gene alteration status are required to be collected and documented to determine the eligibility of the study. For the Phase II stage, besides the local laboratory test results of MAPK pathway gene alteration status, a molecular screening assessing archival and/or fresh FFPE tumor samples is mandatory for a confirmatory detection of MAPK pathway gene status by a Sponsor designated central laboratory.

MAPK pathway genetic alteration status information collected before taking part in study might be acceptable, if already documented in your medical records.

Potential biomarkers for HH2710 response or resistance in blood or tumor specimens, including but not limited to genetic alterations in the MAPK pathway, will also be studied.

Molecular screening testing can be done while you are receiving standard treatment for your tumor or whenever possible.

#### **Procedures**

Tumor biopsy or tissue samples will be collected for molecular screening.

Your samples will be coded before being shipped to a Sponsor designated central laboratory and will be stored there until they are analyzed. Staff members there are experienced in handling and testing samples from research studies.

Your samples will only be used for study-related purposes. No other analyses will be performed without your approval and the approval of the Ethics Committee. You have the right to refuse permission for these additional tests to be done, and you may (at any time) request that your samples be destroyed.

You may also request that all previously retained samples be destroyed. Your samples will not be used for any new tests, however, the information already gathered from your samples will be retained for the integrity of the study.

### Risks and discomforts

"Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inVentiv Health group of companies"


Principal Investigator: <PI name>; Site No.: <site #>

The risks of a biopsy can include bleeding, pain, and infection. To reduce these risks, the site of the biopsy will be numbed and sterile techniques will be used.

When your blood is drawn, you may feel light-headed. At the site where the blood was drawn, you may have inflammation of the vein (blood vessel), pain, bruising, or bleeding. There is also a low possibility of infection.

### Confidentiality and data protection

Information provided in the main informed consent form in Appendix 1 (Privacy Notice) applies for this testing. Your identity will not be disclosed unless required by law.

### **Insurance**

Information provided in the main subject information sheet and informed consent form in the "What if I get sick or hurt" section applies for this testing.

### Compensation

You will not have to pay to take part in this testing, and you will not be paid for your participation in this testing. If the Sponsor is able to create or design new tests or medications as a result of this study, you will not receive any money (reimbursement) because of your participation in this testing.

### **Potential benefit**

Being in the sub-studies will not directly help you. Information from the sub-studies may help researchers understand advanced tumors, respond to treatment, and discover new tests or medications to help patients with this disease, possibly including you, in the future.

### **Voluntary participation and withdrawal**

Your participation in this testing is voluntary. You do not have to take part in this testing if you do not want to take part. In case you refuse to participate in this analysis, you cannot participate in the main study in Phase II stage.

If you do not want to take part in this sub-study, there will be no penalty to you. You will not lose any benefits to which you are otherwise entitled, and your regular medical care at this study site will not change.

You can stop your participation in this testing at any time without giving any reason by informing your study doctor. Your samples will be destroyed, and no new data will be collected about you after you withdraw from this testing.

### **Contact person**


Principal Investigator: <PI name>; Site No.: <site #>

If you have any questions about this testing, please contact the study doctor, Dr [name of principal investigator] at [phone number] or [name of sub-investigator, research nurse, etc] at [phone number].


Principal Investigator: <PI name>; Site No.: <site #>

# **Consent to Participate**

By signing this informed consent form, I agree to the following:

- I have read and I understand this informed consent form.
- I confirm that the substudy has been explained to me.
- I have been given the chance to ask questions that I have had about this testing, and all questions that I have asked have been answered to my satisfaction.
- I know who to contact if I have any further questions.
- I confirm that I voluntarily agree to participate in this testing.

| An original | copy of the | information | sheet and | signed | consent | form | will b | e given | to you | u to |
|---|---|---|---|---|---|---|---|---|---|---|
| keep. | | | | | | | | | | |

| Name of participant (print) | |
|---|---|
| Signature of participant | Date (dd/Mmm/yyyy) |
| Signature of study doctor or person administering consent | Date (dd/Mmm/yyyy) |

<sup>&</sup>quot;Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inVentiv Health group of companies"

ClinicalTrials.gov ID: NCT04198818

**Pregnant Partner Informed Consent Form** 


Principal Investigator: <PI name>; Site No.: <site #>

# **Pregnant Partner Informed Consent Form**

**Study Title:** A First-in-Human, Open Label, Phase I/II Study to Evaluate the Safety,

Tolerability and Pharmacokinetics of HH2710 in Patients with Advanced

**Tumors** 

**Protocol Number:** HH2710-G101

**Sponsor:** Haihe Biopharma Co., Ltd.

Name of Doctor or Other Person Administering Consent: [Name of doctor/other person]

Principal Investigator: [Insert name, affiliation, location]

Telephone number:

Daytime: [Phone number]

After office hours: [After hours phone number]

# **Introduction and Purpose of the Form**

Your partner, the biological father of your baby, is/was participating in the clinical trial listed above, whose primary purpose is/was to learn how well the study drug works and how safe the study drug (HH2710) is for treating patients with advanced tumors.

You have become pregnant while your partner is/was taking part in this clinical study or in the 6 months after he discontinued from the study drug.

As the effect and risks of the study drug on sperm, ova, unborn children, and infants are not known, we kindly request that you sign this consent form to allow the collection of data related to your and your baby's health conditions both during your pregnancy and after the outcome of your pregnancy.

The data collected will only be processed to the extent necessary to monitor the health of you and your baby during your pregnancy and potentially after the outcome of your pregnancy. Data collected will help doctors monitor the potential risks to you or your baby as a result of your partner's exposure to the study drug.

The data will be collected by the study doctor for reporting of side effects.

Please take time to read the following information. Your participation in this data collection research is voluntary. You do not have to agree to have information about your pregnancy collected, and you can change your mind at any time. If you do not agree to have information about your pregnancy collected, this will not affect your partner's ability to participate in the

Pregnant Partner ICF Version Number: 2.1 Date: 18-Feb-2021 Controlled Document ID: **4106B.00**, Effective Date: 30-Apr-2018


Principal Investigator: <PI name>; Site No.: <site #>

research study. Your decision will not affect you, your partner's, or your baby's regular medical care.

### Type of information requested

With this form, we are asking for your permission to collect medical information about your pregnancy, its outcome, the date of conception, medications/medical treatments that you have taken/received or may take/receive during your pregnancy, and, if appropriate, information about the birth and health of your baby (including sex, birth weight, and size), as well as information about your personal health, now and in the past, including information on prior pregnancies, if any. The goal of this data collection is to determine if the study drug that your partner was given has an effect on your pregnancy and/or the health of your baby. Also, your demographic data and personal data on your physical or disease condition may be collected. Your identity and that of your baby, however, will be kept secret and will not be collected.

This information will be collected, if appropriate, until your baby is born.

# Possible side effects, risks, or discomforts

The study doctor will not perform any examinations, tests, or procedures on you.

Your only involvement in the study will be to answer questions and provide information.

### **Benefits**

There are no direct benefits to you or your baby for agreeing to share your data. However, we hope that the information we gather about your pregnancy will help future patients and their partners by helping us understand the potential risks of the study drug.

### Compensation

You will not be paid for the collection of your and your baby's personal and health data.

### **Confidentiality and data protection**

For your data to be used, you must read and sign the Privacy Notice at the end of this form (see Appendix 1).

### **Insurance**

You should contact your health insurance to understand your coverage.

### Contact person

For safety reasons, it is recommended that your general practitioner, obstetrician or gynecologist, or other specialist is informed about your pregnancy and that your partner is taking part in a research study.

<sup>&</sup>quot;Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inVentiv Health group of companies"


Principal Investigator: <PI name>; Site No.: <site #>

If you have any questions about this form or how your information will be used, please contact your partner's study doctor at the address and/or telephone number provided below. The study doctor is collecting only information related to the progress of your pregnancy and its outcome; you should contact your regular health care providers for any health concerns that you may have.

<Insert address and contact information of study doctor.>

### **Authorization for Release of Medical Information**

Study Title: A First-in-Human, Open Label, Phase I/II Study to Evaluate the Safety, Tolerability

and Pharmacokinetics of HH2710 in Patients with Advanced Tumors

**Protocol Number:** HH2710-G101 **Sponsor:** Haihe Biopharma Co., Ltd.

Principal Investigator: [Insert name, affiliation, location]

Telephone number:

Daytime: [Phone number]

After office hours: [After hours office number]

- I have read, and I understand the information provided in this form.
- I have been given the chance to ask questions that I have had about the study, and all questions that I asked have been answered to my satisfaction.
- I understand that I will not receive any benefits from providing my and my baby's health information.
- I freely consent to allow the use and disclosure of my and my baby's health information in connection with this safety activity as described in this Authorization Form.
- I understand that I am free to withdraw my consent at any time for any reason. I will tell the study doctor if I decide to withdraw my consent.
- I consent to provide the contact data of my pregnancy healthcare provider to my partner's study doctor.
- I understand that I will receive a signed and dated copy of this Authorization Form for my records.

My consent to participate in this study does not take away any legal rights in the case of negligence (carelessness) or other legal fault of anyone who is involved with this study.

<sup>&</sup>quot;Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inVentiv Health group of companies"

Pregnant Partner Informed Consent Form
Principal Investigator: <PI name>; Site No.: <site #>

| Read and understood | |
|---|---|
| Pregnant Partner's first and last name (Print) | |
| Signature of Pregnant Partner | Date (dd/Mmm/yyyy) |
| Subject's first and last name and study ID number (Print) | |
| Signature of study doctor or person administering consent | Date (dd/Mmm/yyyy) |

"Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inVentiv Health group of companies"


Principal Investigator: <PI name>; Site No.: <site #>

Appendix 1: Privacy Notice

**Identification of Data Controller:** During the study, the Sponsor will direct the collection and use of your personal information (data) needed for the outcome of your pregnancy. The Sponsor is the data controller of your and your baby's personal data under applicable data protection laws. You can contact the Sponsor at:

Ms. Xianqing Hu

No. 865 Zuchongzhi Road, Pudong New Area, Shanghai, China

Tel: +86 21 20568888

The study center may also be considered as a data controller of your and your baby's personal data under applicable data protection laws. You may contact the study doctor using the contact information for the study doctor on the first page of this informed consent form. <a href="#style="contact: 150%;">If relevant> You can contact the study center's data protection officer at: 55tudy center to provide contact information></a>.

If you have any questions or would like to see the data collected about you and your baby for this study, you should contact the study doctor.

**Data to be Collected and Processed:** The study staff will collect health information about you and your baby. This data may include your name or initials, date of birth, gender, and contact details and information about the birth and health of your baby such as sex, birth weight, and size. In addition, the following sensitive personal data about you may be collected: health, ethnicity, race, sexual activity or orientation, genetic information, and fingerprints or eye scans (to help verify your identity).

How Your and Your Baby's Personal Data Will be Used: The personal data collected about you and your baby will be recorded in your partner's study file by the study staff to monitor your and your baby's safety. Your and your baby's personal data may be processed on a computer and/or on paper. The collection of this data is necessary to determine if the study drug that your partner was given has an effect on your pregnancy and/or the health of your baby.

There are laws about the recording, forwarding, storage, and analysis of your and your baby's personal data, including sensitive personal data. These laws require your voluntary and explicit consent before any data are collected about you and your baby.

Results of this study may be presented at meetings or in publications; however, your identity will never be shared. Your personal data will not be used for any direct marketing purposes.

If information regarding a communicable disease is collected, the information may be shared with a public health authority that is authorized by law to collect or receive such information for

<sup>&</sup>quot;Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inVentiv Health group of companies"


Principal Investigator: <PI name>; Site No.: <site #>

the purpose of preventing or controlling disease, injury, or disability, and conducting public health surveillance, investigations, or interventions.

**Storage of Your and Your Baby's Personal Data:** According to legal requirements, your personal data will be stored in the study databases and/or paper files for at least 15 years after the study ends, as required by applicable laws.

Transferring the Personal Data to a Third Party: To keep your and your baby's identity private, all data that is sent or provided outside of the study center will show only a coded identification number instead of your name. Only the study doctor and authorized personnel will be able to connect this code to your name. They will use a list that will be kept in a secure place to link this code to your name in case of an emergency. The coded data from the study showing your and your baby's involvement (including uncoded personal information) will be provided to the Sponsor and other individuals and/or companies that act on the Sponsor's behalf, including Syneos Health. Also, your and your baby's medical records (including uncoded personal data) may be reviewed by the Sponsor and other individuals and/or companies that act on the Sponsor's behalf, including Syneos Health; government agencies in countries where the study drug may be considered for approval (such as the US FDA); [IRB/IEC name], a group that reviews and approves studies; and independent auditors for the purposes of monitoring your and your baby's safety. Further, your and your baby's personal information may be disclosed in response to lawful requests by public authorities, including those to meet national security or law enforcement requirements.

If your and your baby's personal data is shared with other companies that are located outside of the country where you live, the Sponsor will make sure that your and your baby's data is protected as required by your country's data protection laws. Some of these other companies may be located in countries whose data protection and privacy laws may be less strict than in your own country, including the United States and \_\_\_\_\_\_\_. You may contact the study doctor to get more information about the precautions used to protect your and your baby's personal data outside of your country. You may also ask the study doctor for a copy of those precautions.

With your permission, the study doctor will tell your primary doctor about your role in this study.

A description of this clinical trial will be available on http://www.clinicaltrials.gov as required by US law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

Your Rights as a Data Subject: You have the right to access and correct the data collected about you and your baby during the study and submit any questions or concerns about the collection or processing of your and your baby's personal data, however this access is suspended until after the study has ended. Your rights will be reinstated at the conclusion of the study.

<sup>&</sup>quot;Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inVentiv Health group of companies"


Principal Investigator: <PI name>; Site No.: <site #>

You may make these requests by contacting the study doctor. You may also have the right to file a complaint regarding the handling of your and your baby's personal information with your local data protection authority.

You have the right to withdraw your consent for the processing of your and your baby's personal data at any time. You must withdraw your consent by writing to the study doctor. However, data collected before you remove your consent is still legally allowed to be used.

### Consent Language

### Consent to the Collection, Processing, and Use of Personal Data

By signing below, I agree that:

- (1) My and my baby's personal data, including sensitive personal data, can be collected, used, and archived for purposes of determining if the study drug my partner was given has any effect on my pregnancy and/or the health of my baby as described in this Privacy Notice
- (2) My and my baby's personal data, including sensitive personal data, can be transferred to and shared with other companies both within and outside of the European Economic Area (EEA), including to countries that may not have the same level of data protection as the EEA, as described in the Privacy Notice

This consent is valid unless you change your mind and provide a written notice to the study doctor. You will receive a signed and dated copy of this Privacy Notice.

| Pregnant Partner's First and Last Name (print) | |
|---|---|
| Signature of Pregnant Partner | Date (dd/Mmm/yyyy) |
| Subject's First and Last Name and Study ID number (Print) | |

<sup>&</sup>quot;Syneos Health" as used in this document includes Syneos Health, Inc. and its operating companies and subsidiaries which include but are not limited to the INC Research group of companies and the inVentiv Health group of companies"